CLINICAL TRIAL: NCT01600521
Title: A Clinical Study of a Natural Remedy for Rheumatoid Arthritis vs. Commonly Used Conventional Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1205E14290
Record Dates: First submitted 2012-04-05; First posted 2012-05-17 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paeoniflorin + Polypeptides (PAE + CCPI) (Active Comparator): Paeoniflorin (PAE), the extract from peony (Paeonia lactiflora), is an active ingredient with anti-inflammation properties. Polypeptides (3,000 - 10,000 dalton) in Cervus & Cucumis polypeptide injection (CCPI), the extract from Sika deer (Cervus nippon Temmick) bones and muskmelon (Cucumis melo L) seeds, are the active ingredients with bone healing, pain relieving, and anti-inflammation properties. PAE was administrated orally 600 mg twice a day for at least 12 months. CCPI was administered intravenously 8~12 mL daily with 250 mL 5% dextrose injection solution or 0.9% NaCl IV solution for 2 weeks, discontinued 1 week, and restarted for another 2 weeks.
  Interventions: Drug: A Natural Remedy for Rheumatoid Arthritis vs. Common Drugs
- Methotrexate (MTX) + Leflunomide (LEF) (Active Comparator): DMARDs (methotrexate: MTX, leflunomide: LEF) were taken orally for at least 12 months. MTX dose: 7.5 mg ~ 10mg / week, LEF dose: 10 mg ~ 20mg daily.
  Interventions: Drug: A Natural Remedy for Rheumatoid Arthritis vs. Common Drugs
- MTX + LEF + CCPI (Active Comparator): The DMARDs and CCPI were administrated as in the above two groups.
  Interventions: Drug: A Natural Remedy for Rheumatoid Arthritis vs. Common Drugs

INTERVENTIONS:
Drug: A Natural Remedy for Rheumatoid Arthritis vs. Common Drugs — The comparisons of the efficacy and safety of the following treatments for rheumatoid arthritis: paeoniflorin (PAE) + Cervus and Cucumis polypeptide injection (CCPI), methotrexate (MTX) + leflunomide (LEF), and MTX + LEF + CCPI.
  Other Names: TGP: Lansen Pharmaceuticals, China. Brand name: Pafulin.; CCPI: Gloria Pharmaceuticals, China. Brand name: Songmeile.; MTX: Shanghai Sine Pharmaceuticalx, China.; LEF: Changzheng-Xinkai Sino-American Pharmaceutical, China

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a combined therapy for rheumatoid arthritis (RA). The combined therapy contained paeoniflorin (Brand name: Pafulin), which has anti-inflammation properties, and Cervus and Cucumis polypeptide injection (Brand name: Songmeile), which has bone healing, pain relieving, and anti-inflammation properties. The hypothesis is that this remedy, which has long been used by the world's largest RA community, is effective and safe when tested by modern clinical standards and criteria.

DETAILED DESCRIPTION:
This is a double-blinded randomized study on the treatment of rheumatoid arthritis. In particular, patients were randomly assigned to one of the following treatment groups: Paeoniflorin (PAE) + Cervus and Cucumis polypeptide injection (CCPI), Methotrexate (MTX) + Leflunomide (LEF), and MTX + LEF + CCPI. The therapeutic effectiveness was evaluated by the 7 core set measures of American College of Rheumatology (ACR). Adverse effects, their severity, and the evaluators' professional judgments of relationships between the adverse effects and the drugs were documented.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or older
* active RA, defined by at least 8 swollen joints and at least 10 tender joints (excluding distal interphalangeal joints)
* an erythrocyte sedimentation rate (ESR) of at least 28 mm per hour
* the 1987 revised American College of Rheumatology (ACR) criteria for diagnosis of RA for at least 6 months
* not use of NSAIDs within two weeks
* agreement to participate in this study.

Exclusion Criteria:

* poor compliance
* severe medical conditions
* abnormalities in liver, or kidney function, or in haematological parameters,
* pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1748 (Actual)
Dates: Start 2004-11; Primary Completion 2011-04 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The relief of rheumatoid arthritis symptoms and the improvement of functions assessed by the American College of Rheumatology (ACR) core set measures. | CCPI: 2 weeks + 2 weeks with 1 week in between. All other drugs: at least 12 months.
  The American College of Rheumatology (ACR) core set measure improvement % response rate was used to assess the relief of rheumatoid arthritis symptoms and the improvement of functions.

SECONDARY OUTCOMES:
The adverse effects associated with the treatments | CCPI: 2 weeks + 2 weeks with 1 week in between. All other drugs: at least 12 months.
  The following parameters were used to measure the safety of the treatments: Headache, Up resp infection, Urinary tract infection, Other infection, Nausea, Rash, Diarrhea, Fatigue, Alopecia, Rhinitis, Dizziness, Abdominal pain, Sinusitis, Mouth ulcer, Hypertension, Dyspepsia, Vomiting, Insomnia, ALT elevation, AST elevation, WBC decrease, Glucose elevation, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Affiliated to Capital Medical University, Beijing
  - Institute of Chinese Medical Sciences, University of Macau, Taipa

REFERENCES:
- [Derived] Chen L, Qi H, Jiang D, Wang R, Chen A, Yan Z, Xiao J. The new use of an ancient remedy: a double-blinded randomized study on the treatment of rheumatoid arthritis. Am J Chin Med. 2013;41(2):263-80. doi: 10.1142/S0192415X13500195. PMID 23548118
- See also: China has the world's largest RA patient population. Its population is more than four times the population of the United States (1,346vs.312 millions), and almost two times the total populations of all European countries combined (1,346vs.740 millions) — http://www.prb.org/pdf11/2011population-data-sheet_eng.pdf